CLINICAL TRIAL: NCT04422834
Title: The Reliability, Validity and Cross-Cultural Adaptation of the Turkish Version of Jefferson Scale of Empathy For Health Professional Students
Brief Title: Translation and Validation of the Turkish Version of JSE-HPS
Acronym: JSE-HPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Alper Tuğral, Alper Tuğral, Izmir Bakircay University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BakircayU07/07022020
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Surveys and Questionnaires; Empathy
Keywords: Jefferson Scale of Empathy; Empathy; Questionnaire
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: A group of students who studying at Faculty of Health Sciences will be asked to fill Turkish version of JSE-HPS and ETS. JSE-HPS will be asked to re-fill after seven days for retest analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Professional Students (Experimental): A group of students who studying at the Faculty of Health Sciences will be asked to fill the Turkish version of JSE-HPS and ETS. JSE-HPS will be asked to re-fill after seven days for retest analysis.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A group of students who studying at the Faculty of Health Sciences will be asked to fill the Turkish version of JSE-HPS and ETS. JSE-HPS will be asked to re-fill after seven days for retest analysis.

SUMMARY:
Empathy, which can be briefly defined as understanding and feeling of one's thoughts upon experiences. It has been gaining importance in health care. A great majority of the literature has been focusing on the aspect of physician and health care provider yet recently establishing or measuring empathy has been performed with the undergraduate students. Since empathy and its related dimensions are important to integrate a better skill to provide in health care, measuring empathy gained attention. However, there might be lacking some tools which assess empathy directly such as the Empathic Tendency Scale and the Empathic Skill Scale in the Turkish language, yet these were discussed as cannot be quite modifiable to some specific sub-groups such as health sciences students. Thus, this study is aimed to study for the reliability, validity, and cross-cultural adaptation of the Turkish version of the Jefferson Scale of Empathy for undergraduate health care students.

DETAILED DESCRIPTION:
The research has been aimed at studying translation, validation, a cross-cultural adaptation of the Turkish version of the Jefferson Scale of Empathy for Health Professional Students (JSE-HPS).

Study Setting:

This research was planned as a descriptive study. The research is planning to be performed between May 2020 and October 2020. The students who are currently studying in the Faculty of Health Sciences will be asked to participate in this study. Since ethical board approval was taken in February 2020 and study was planned to start in March or April 2020. However, due to the Covid-19 pandemic, the research in which test and re-test protocols should be performed by students was re-planned by doing these protocols via internet-based forms. Before the study, all participating students were informed about this study. To achieve their consent in regard to participate in this study, a "tick-box" was placed prior to the questionnaire in which whether they accept that participating in this study voluntarily. The primary target for sample size was set as 300 students.

Measurement and Method:

The descriptive data will be gathered by using the Jefferson Scale of Empathy for health professional students (JSE-HPS), the Turkish version of Empathic tendency scale (ETS), and sociodemographic form in which age, gender, and other information will be requested to fill out.

JSE-HPS:

JSE-HPS was originally developed by Jefferson University. It consists of 20 items each scored according to the seven-point Likert type scale in which 1 means "Strongly Disagree" while 7 means "Strongly agree". The minimum and maximum scores range from 20 to 140. Higher scores indicate a better empathic aspect or vice versa.

Empathic Tendency Scale (ETS):

ETS was originally developed in the Turkish language in 1988. Turkish validation and reliability of ETS were also conducted and found to reliable according to the Cronbach's alpha value is 0.82. ETS consists of 20 items each scored according to the five-point Likert type scale in which 1 equals "Completely contradictory" while 5 means "Completely proper". Each item is related to some ideas which are quite common in daily life. 20 and 100 are minimum and maximum scores, respectively. Higher scores indicate a better empathic aspect.

Translation and Cross-cultural Adaptation Process:

The permission was granted from the copyright Holder of JSE-HPS in order to study the reliability, validity, and adaptation of the Turkish version of JSE-HPS. The cultural adaptation was performed according to the protocol explained by Beaton et al. Steps and a detailed explanation of this protocol can be found in the literature. Briefly, an expert committee consists of study researchers separately translated the original version of the JSE-HPS into Turkish. The final version of the Turkish translated JSE-HPS was created according to the separately translated ones. This final version was re-translated to English by a native English speaker who is also capable to talk Turkish language. The expert committee eventually made a final version to which can be applicable to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Being currently studying at the Faculty of Health Sciences
* Able to read, write and understand the Turkish language
* Having no mental medical conditions
* Being a volunteer to participate in this study

Exclusion Criteria:

* Inability to read, write and understand Turkish language
* Not volunteer to participate in this study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Jefferson Scale of Empathy Health Professional Students Questionnaire | Baseline
  The Turkish version of Jefferson Scale of Empathy Health Professional Students (JSE-HPS) will be applied to participants. The minimum and maximum scores for JSE-HPS can be reached to 20 and 140, respectively. The more the higher scores indicate more empathic aspect or vice versa.
Jefferson Scale of Empathy Health Professional Students Questionnaire | 1 week after baseline
  The Turkish version of Jefferson Scale of Empathy Health Professional Students (JSE-HPS) will be applied to participants. The minimum and maximum scores for JSE-HPS can be reached to 20 and 140, respectively. The more the higher scores indicate more empathic aspect or vice versa.
Empathic Tendency Scale (ETS) Questionnaire | Baseline
  The Turkish version of Empathic Tendency Scale (ETS) Questionnaire will be applied to participants. The minimum and maximum scores can be taken from the tool are 20 and 100, respectively in which higher scores indicate better empathic attitude or vice versa.

SECONDARY OUTCOMES:
Demographic Data Form | Baseline
  Basic Form gathers some information related participants' age, gender etc.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Günay İsmailoğlu, PhD, Principal Investigator — Izmir Bakircay University; Kadirhan Özdemir, PhD, Principal Investigator — Izmir Bakircay University
Locations (1):
- İzmir Bakırçay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anfossi M, Numico G. Empathy in the doctor-patient relationship. J Clin Oncol. 2004 Jun 1;22(11):2258-9; author reply 2259-60. doi: 10.1200/JCO.2004.99.302. No abstract available. PMID 15169824
- [Background] Hojat M, Louis DZ, Markham FW, Wender R, Rabinowitz C, Gonnella JS. Physicians' empathy and clinical outcomes for diabetic patients. Acad Med. 2011 Mar;86(3):359-64. doi: 10.1097/ACM.0b013e3182086fe1. PMID 21248604
- [Background] Kim SS, Kaplowitz S, Johnston MV. The effects of physician empathy on patient satisfaction and compliance. Eval Health Prof. 2004 Sep;27(3):237-51. doi: 10.1177/0163278704267037. PMID 15312283
- [Background] Hogan R. Development of an empathy scale. J Consult Clin Psychol. 1969 Jun;33(3):307-16. doi: 10.1037/h0027580. No abstract available. PMID 4389335
- [Background] Fields SK, Hojat M, Gonnella JS, Mangione S, Kane G, Magee M. Comparisons of nurses and physicians on an operational measure of empathy. Eval Health Prof. 2004 Mar;27(1):80-94. doi: 10.1177/0163278703261206. PMID 14994561
- [Background] Sherman JJ, Cramer A. Measurement of changes in empathy during dental school. J Dent Educ. 2005 Mar;69(3):338-45. PMID 15749944
- [Background] Fields SK, Mahan P, Tillman P, Harris J, Maxwell K, Hojat M. Measuring empathy in healthcare profession students using the Jefferson Scale of Physician Empathy: health provider--student version. J Interprof Care. 2011 Jul;25(4):287-93. doi: 10.3109/13561820.2011.566648. Epub 2011 May 9. PMID 21554061